CLINICAL TRIAL: NCT05852197
Title: Effect of Anticoagulant Drug Intervention on postoperativeMajor Adverse Limb Events and Major Adverse Cardiovascular Events in Patients With Peripheral Arterial Disease
Brief Title: Effect of Anticoagulant Drug Intervention on Postoperative MALE and MACE in Patients With PAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20230084B
Record Dates: First submitted 2023-04-22; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-02

CONDITIONS: Anticoagulant Drugs; Antiplatelet Drug; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Anticoagulants; Platelet Aggregation Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Use a combination of anticoagulant or antiplatelet drugs ， group 1
  Interventions: Drug: anticoagulant or antiplatelet drugs
- Use a combination of anticoagulant or antiplatelet drugs， group 2
  Interventions: Drug: anticoagulant or antiplatelet drugs

INTERVENTIONS:
Drug: anticoagulant or antiplatelet drugs — combination of anticoagulant or antiplatelet drugs

SUMMARY:
Patients with PAD were grouped according to the combination of different anticoagulant and antiplate drugs. The type, dosage and duration of anticoagulant and antiplatelet drugs were recorded after operation. Major Adverse Cardiovascular Events and Major Adverse Limb Events were followed up at 1 month, 6 months and 12 months, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years old
2. Patients with symptomatic PAD
3. Moderate intermittent claudication, or severe limb ischemia
4. Radiographically confirmed occlusion
5. Received a successful revascularization

Exclusion Criteria:

1. Acute limb ischemia occurred within 2 weeks before revascularization;
2. Large tissue defect of any lower limb (defined as obvious ulceration/gangrene near phalangeal head);
3. After revascularization, there are clinical conditions requiring systemic anticoagulation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intracavitary therapy for lower extremity arteriosclerosis obliterans
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite adverse event incidence (MACE/MALE) : myocardial infarction, ischemic stroke, acute limb ischemia, major amputation due to vascular disease | The 1st month after treatment
  The incidence of myocardial infarction, ischemic stroke, acute limb ischemia, and major amputation owing to vascular disease after the treatment. Measured in the first, sixth, ninth, and twelfth month.
Composite adverse event incidence (MACE/MALE) : myocardial infarction, ischemic stroke, acute limb ischemia, major amputation due to vascular disease | The 3rd month after treatment
  The incidence of myocardial infarction, ischemic stroke, acute limb ischemia, and major amputation owing to vascular disease after the treatment. Measured in the first, sixth, ninth, and twelfth month.
Composite adverse event incidence (MACE/MALE) : myocardial infarction, ischemic stroke, acute limb ischemia, major amputation due to vascular disease | The 6th month after treatment
  The incidence of myocardial infarction, ischemic stroke, acute limb ischemia, and major amputation owing to vascular disease after the treatment. Measured in the first, sixth, ninth, and twelfth month.
Composite adverse event incidence (MACE/MALE) : myocardial infarction, ischemic stroke, acute limb ischemia, major amputation due to vascular disease | The 9th month after treatment
  The incidence of myocardial infarction, ischemic stroke, acute limb ischemia, and major amputation owing to vascular disease after the treatment. Measured in the first, sixth, ninth, and twelfth month.
Composite adverse event incidence (MACE/MALE) : myocardial infarction, ischemic stroke, acute limb ischemia, major amputation due to vascular disease | The 12th month after treatment
  The incidence of myocardial infarction, ischemic stroke, acute limb ischemia, and major amputation owing to vascular disease after the treatment. Measured in the first, sixth, ninth, and twelfth month.

SECONDARY OUTCOMES:
MACE | The 1st，3rd，6th，9th，12th month
  The incidence of myocardial infarction, ischemic stroke owing to vascular disease after the treatment. Measured in the first, sixth, ninth, and twelfth month.
MALE | The 1st，3rd，6th，9th，12th month
  The incidence of acute limb ischemia, major amputation due to vascular disease owing to vascular disease after the treatment. Measured in the first, sixth, ninth, and twelfth month.
Compound protection from vasogenic adverse events | The 1st，3rd，6th，9th，12th month
  The incidence of muscle infarction, ischemic stroke, acute limb ischemia, major amputation due to vascular disease, massive bleeding after the treatment. Measured in the first, sixth, ninth, and twelfth month.
all-cause mortality | The 1st，3rd，6th，9th，12th month
  Deaths occurring during follow-up, regardless of cause
health economics evaluation | The 1st，3rd，6th，9th，12th month
  The cost of patient treatment

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, None Selected, China

IPD SHARING:
Plan to Share IPD: Yes
With the consent of the committee, it can be based on patient data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code